CLINICAL TRIAL: NCT01884363
Title: Walnut Consumption, Endothelial Function, and Plasma Adipokines in Subjects With Diabetes or Coronary Disease: a Pilot Trial
Brief Title: Walnut Consumption, Endothelial Function, and Biomarkers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Luc Djousse, Director of Research, Associate Professor of Medicine, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: 2013P000803
Record Dates: First submitted 2013-06-19; First posted 2013-06-24 (Estimated); Last update posted 2016-03-18 (Estimated); Status verified 2016-03

CONDITIONS: Coronary Heart Disease; Type 2 Diabetes
Keywords: Endothelial function; walnuts; clinical trial; Nutrition; cardiovascular disease
MeSH Terms: conditions — Coronary Disease; Diabetes Mellitus, Type 2; Cardiovascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Walnuts (Experimental): This group will receive one ounce of walnuts per day
  Interventions: Other: Once ounce per day of walnuts
- Usual diet (no walnuts) (No Intervention): Control group (does not receive walnuts in the diet)

INTERVENTIONS:
Other: Once ounce per day of walnuts
  Arms: Walnuts

SUMMARY:
This study will examine whether a twelve-week intervention with one ounce (28 g) per day of walnuts improves endothelial function measured non-invasively using finger probe (EndoPat-2000) in people with coronary heart disease or type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Age 30+ years
* Prevalent coronary artery disease
* Prevalent type 2 diabetes

Exclusion Criteria:

* Current eating disorder
* Pregnant or lactating women
* Allergy to walnuts or other nuts
* Inability to provide informed consent or blood samples
* History or prevalent diagnosis of cancer, asthma, kidney insufficiency, stroke, seizures, allergic disorders, or congestive heart failure
* Diagnosis of coronary heart disease or diabetes < 1 year prior to enrollment
* Intention to move out of greater Boston area within one year
* Current use of walnuts for more than 2 ounces per day
* Bleeding disorder
* Treatment with blood thinning drugs (i.e. warfarin, clopidogrel)
* Major surgical operation 3 months before or after screening
* Organ transplantation
* Current participation in another trial or plan to do so during the study
* Use of vasodilators such as nitroglycerin
* Inability to give informed consent
* Inability to travel to the study center at Brigham and Women's Hospital

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2013-06; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Change in reactive hyperemia index occurring between baseline and 12 weeks (end of intervention) | 12 weeks
  Reactive hyperemia index (RHI), which in part reflects vasodilator function of the small blood vessel at the fingertips is an indirect measure of endothelial function. Change in RHI between baseline and 12 weeks post intervention will be measured in each group using EndoPat2000 device. We will compare RHI change between walnut group and usual diet group.

SECONDARY OUTCOMES:
Change in blood levels of hormones produced by fat cells between baseline and 12 weeks (end of intervention) | 12 weeks
  Specifically, we will measure changes in blood levels of following hormones: retinol binding protein 4, fatty acid binding protein 4, total adiponectin, and leptin before and after 12 weeks of walnut consumption/consumption of usual diet.

OTHER OUTCOMES:
Change in heart rate variability between baseline and 12 weeks post-intervention | 12 weeks
  Change in heart rate variability will be measured in each group before and after 12 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Luc Djousse, MD, ScD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Background] Djousse L, Lu B, Gaziano JM. Effects of Walnut Consumption on Endothelial Function in People with Type 2 Diabetes: a Randomized Pilot Trial. Curr Nutr Rep 2016;5:1-8